CLINICAL TRIAL: NCT03752892
Title: Randomized Controlled Trial of Partitioned Aerobic Exercise Training of Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Partitioned Training of Patients With Idiopathic Pulmonary Fibrosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Director, Program in Respiratory Rehabilitation, West Park Healthcare Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1L-IPF-RCT-RG2018
Record Dates: First submitted 2018-11-20; First posted 2018-11-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lung; Disease, Interstitial, With Fibrosis
Keywords: pulmonary rehabilitation; exercise training
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: prospective, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: assessor of the primary outcomes will be blind to the participant's group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention -1-leg cycle training (Experimental): Primary aerobic training component one-legged, partitioned, cycle training. A progressive approach to combined intensity and duration will be taken. A cycle starting with intermittent high intensity one-legged exercise progressing to continuous duration of the target duration of 15 min for each leg and then restarting the cycle at a higher intensity.
  Interventions: Other: intervention -1-leg cycle training
- usual care - 2-leg cycle training (Active Comparator): Primary aerobic training component conventional two-legged cycle training. A progressive approach to combined intensity and duration will be taken. A cycle starting with intermittent high intensity exercise progressing to continuous duration of 30 min and then restarting the cycle at a higher intensity.
  Interventions: Other: usual care - 2-leg cycle training

INTERVENTIONS:
Other: intervention -1-leg cycle training — partitioned aerobic exercise training
  Arms: intervention -1-leg cycle training
Other: usual care - 2-leg cycle training — conventional aerobic exercise training
  Arms: usual care - 2-leg cycle training

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a lung disease that limits the ability to breathe enough for a good workout. One way to improve the exercise training is to reduce the number of muscles being trained together. By training one leg at a time, the patient does not have to breathe as much allowing each leg a better workout. Our groundwork suggests it may work in patients with IPF. This study will help decide whether one-legged exercise training is better at improving a patient's exercise endurance compared to the usual way of exercising with both legs at the same time.

DETAILED DESCRIPTION:
Dyspnea is a major clinical manifestation of idiopathic pulmonary fibrosis (IPF). It becomes more severe and more limiting as the condition progresses. Many professional respiratory societies recommend that the standard of care for IPF includes pulmonary rehabilitation (PR). However, some patients with IPF are so limited by dyspnea that they are unable to tolerate levels of aerobic exercise training sufficient to induce the physiological adaptations that will improve functional and health related outcomes. Therefore, there is a need for exercise training interventions that will enhance the muscle training stimulus above that currently possible in individuals with a marked ventilatory limitation.

Partitioning large muscle exercise using one-legged high intensity training is more effective than conventional aerobic training when applied to patients with central ventilatory or cardiac limitation. Effective partitioned exercise enables an increased muscle load with less ventilatory load. It increases the training stimulus to the muscles as they work at a high intensity, relative to their current aerobic state, necessary to increase their capacity. As long as the active muscle mass can create the same demands on the central exercise components of the heart and circulation as does conventional two-legged exercise, this simple, inexpensive novel approach, will stimulate leg muscles sufficiently to improve overall cardiorespiratory fitness. For example, in those with chronic obstructive pulmonary disease, one-legged training has been shown to provide a muscle specific stimulus sufficient to improve whole body peak oxygen uptake during pulmonary rehabilitation. A preliminary acute study of patients with IPF has demonstrated that during a laboratory simulation of an exercise training session, partitioning aerobic exercise extended exercise tolerance. Participants achieved double the work whilst exercising with one leg compared with two-legged cycle exercise. Partitioned training may therefore be an effective approach to exercise training in patients with IPF enrolled in PR.

The advent of pharmacological agents that stabilize the clinical course of IPF presents a window of opportunity for exercise rehabilitation to further improve function. The aim of this proposed study is to determine whether, within the setting of PR, partitioned aerobic exercise training with a one-legged cycle training regime is more effective than the conventional two-legged regimen in increasing exercise tolerance. The study hypothesis is that partitioned aerobic exercise training, using a one-legged training regime is more effective than conventional two-legged exercise training in increasing exercise tolerance (measured by constant power endurance) and cardiorespiratory fitness as measured by maximal oxygen uptake. The results will inform the best approach to produce clinically meaningful improvements in dyspnea and health status for those with IPF.

ELIGIBILITY:
Inclusion Criteria:

* confirmed idiopathic pulmonary fibrosis
* Clinically stable
* enrolled in pulmonary rehabilitation

Exclusion Criteria:

* co-morbidities that might impair their ability to safely complete a pulmonary rehabilitation program
* complete a pulmonary rehabilitation program within the previous 6 months
* experienced an exacerbation less than six weeks before participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Cycle exercise endurance time | Change from Baseline at discharge from 8 weeks of pulmonary rehabilitation
  tolerance (time) of a constant power high intensity cycle endurance test

SECONDARY OUTCOMES:
health-related quality of life | Change from Baseline at discharge from 8 weeks of pulmonary rehabilitation
  using the questionnaire 'A Tool to Assess Quality of life in IPF' [ATAQ-IPF]

CONTACTS AND LOCATIONS:
Overall Officials: Roger S Goldstein, Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No